CLINICAL TRIAL: NCT03959982
Title: The Effect of Heated, Humidified High-flow Air in COPD Patients With Chronic Bronchitis
Brief Title: HHHFA in COPD Patients, With Chronic Bronchitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spyridon Fortis (Other)
Collaborators: American Thoracic Society (Other)
Responsible Party: Sponsor-Investigator, Spyridon Fortis, Pricipal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201905817
Record Dates: First submitted 2019-05-17; First posted 2019-05-22 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Spirometry; Walking; Tomography, X-Ray Computed

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into two groups: One will receive the device and one will not. Study procedures will be the same for both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HHHFA Randomized Group (Experimental): Subjects will be randomized to use the HHHFA device during bedtime for at least 4 hours. Subjects will complete MRC, SGRQ, CAT, CASA-Q and PSQI questionnaires. They will do spirometry, 6-minute walk, and CT scan. These interventions will be done at baseline and at the completion of their study (6 weeks). Spirehealth Device will be worn by subject daily for 12 weeks.
  Interventions: Device: HHHFA Device; Diagnostic Test: Spirometry; Diagnostic Test: 6-minute walk; Diagnostic Test: CT scan; Other: Medical Research Council dyspnea scale (MRC); Other: St. George's Respiratory Questionnaire (SGRQ); Other: COPD Assessment Test (CAT); Other: Pittsburgh Sleep Quality Index (PSQI); Other: CASA-Q; Other: Spirehealth Tag Device
- Control Group (Active Comparator): Subjects will complete MRC, SGRQ, CAT, and PSQI questionnaires. They will do spirometry, 6-minute walk, and CT scan. These interventions will be done at baseline and at the completion of their study (6 weeks). Spirehealth Device will be worn by subject daily for 12 weeks.
  Interventions: Diagnostic Test: Spirometry; Diagnostic Test: 6-minute walk; Diagnostic Test: CT scan; Other: Medical Research Council dyspnea scale (MRC); Other: St. George's Respiratory Questionnaire (SGRQ); Other: COPD Assessment Test (CAT); Other: Pittsburgh Sleep Quality Index (PSQI); Other: CASA-Q; Other: Spirehealth Tag Device

INTERVENTIONS:
Device: HHHFA Device — Participants will be instructed to use the HHHFA for at least 4 hours during their sleep but will be allowed to use it as long as they want during sleep.
  Arms: HHHFA Randomized Group
Diagnostic Test: Spirometry — Pre and post spirometry using albuterol.
Diagnostic Test: 6-minute walk — 6-minute walk
Diagnostic Test: CT scan — CT scan
Other: Medical Research Council dyspnea scale (MRC) — MRC questionnaire
Other: St. George's Respiratory Questionnaire (SGRQ) — SGRQ questionnaire
Other: COPD Assessment Test (CAT) — CAT questionnaire
Other: Pittsburgh Sleep Quality Index (PSQI) — PSQI questionnaire
Other: CASA-Q — CASA-Q questionnaire
Other: Spirehealth Tag Device — Subjects will wear the Spirehealth Tag Device to measure heart rate, respiratory rate, sleep time, physical activity (movement), and calories burned with activity.

SUMMARY:
Heated, humidified high-flow air (HHHFA) devices improve airway clearance. HHHFA use for an average of 1.6 hours a day in COPD patients with chronic bronchitis improves health-related quality of life, lung function, and delays the first respiratory exacerbation. However, HHHFA for an average of 1.6 hours a day had no effect on COPD exacerbation frequency or hospitalization, dyspnea, or exercise capacity, likely due to short duration of the treatment. Conversely, the effect of HHHFA for longer time periods on chronic bronchitis patients has not been studied. Moreover, the effect of HHHFA on sleep quality has not been studied. A prior study in COPD patients showed that use of HHHFA for more than 7 hours during sleep can be achieved. The overall objective of this research is to examine the effect of HHHFA during sleep on COPD patients with chronic bronchitis. In this pilot study, the study team will examine the effect of HHHFA during sleep on clinically relevant short-term outcomes including: respiratory symptoms, quality of life and sleep, lung function and exercise capacity.

Subjects will be recruited and consented. Once a subject agrees to be in the study the baseline visit will occur. The first test will be the Pulmonary Function testing. If the subject qualifies based on the PFT's they will complete the remainder of the baseline visit. During this visit subjects will complete questionnaires, have a physical, 6 minute walk test and CT scan. Subjects will receive device training on the heated, humidified high-flow air device.

Subjects will have a followup call between 3-7 days to check in on how the subject is doing with the device. After 6 weeks the subject will return for another round of testing as was done at baseline. This will be the final study visit.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is characterized by respiratory exacerbations which increase in frequency as the severity of the disease progresses. COPD exacerbations may lead to hospitalizations, which make up the largest proportion of the total direct health-care cost of the disease and are a significant burden for patients and family. Chronic bronchitis, defined as chronic cough with sputum production for at least 3 months a year for 2 consecutive years, is one of the clinical manifestations of COPD. Chronic bronchitis doubles the risk of COPD exacerbations and hospitalizations, and is associated with increased dyspnea, worse health-related quality of life, and poorer quality of sleep. Chronic bronchitis also results in increased air trapping and hyperinflation, which decreases exercise capacity. Unfortunately, other than traditional inhaled pharmacological agents, there are no treatment options for COPD patients with chronic bronchitis.

Heated, humidified high-flow air (HHHFA) devices improve airway clearance. HHHFA use for an average of 1.6 hours a day in COPD patients with chronic bronchitis improves health-related quality of life, lung function, and delays the first respiratory exacerbation. However, HHHFA for an average of 1.6 hours a day had no effect on COPD exacerbation frequency or hospitalization, dyspnea, or exercise capacity, likely due to short duration of the treatment. Conversely, the effect of HHHFA for longer time periods on chronic bronchitis patients has not been studied. Moreover, the effect of HHHFA on sleep quality has not been studied. A prior study in COPD patients showed that use of HHHFA for more than 7 hours during sleep can be achieved. The overall objective of this research is to examine the effect of HHHFA during sleep on COPD patients with chronic bronchitis. In this pilot study, the study team will examine the effect of HHHFA during sleep on clinically relevant short-term outcomes including: respiratory symptoms, quality of life and sleep, lung function and exercise capacity.

Hypothesis 1: HHHFA during sleep in COPD patients with chronic bronchitis improves respiratory symptoms, sleep quality, lung function, and exercise capacity.

Aim 1: To examine the effect of HHHFA during sleep on respiratory symptoms, sleep quality, lung function, and exercise capacity in COPD patients with chronic bronchitis.

The effect of HHHFA on air trapping and hyperinflation has not been studied. Air trapping and hyperinflation as well as other radiographic measurements associated with chronic bronchitis (e.g. airway wall thickness) can be measured using chest CT.

Hypothesis 2: HHHFA during sleep in COPD patients with chronic bronchitis improves air trapping and hyperinflation.

Aim 2: To examine the effect of HHHFA in COPD patients with chronic bronchitis during sleep on air trapping and hyperinflation through chest CT imaging.

Design: The study team will include COPD subjects with a post-bronchodilator FEV1%predicted below 70% and chronic bronchitis. The study team will include subjects with at least 2 exacerbations in the last year to identify patients with significant burden due to chronic bronchitis. The study team will exclude subjects with recent respiratory events or procedures as the study team want to capture the benefit of HHHFA on chronic, stable COPD participants. Subjects who meet eligibility criteria will be randomized to HHHFA or usual care (Controls). At baseline the study team will perform measurements in all subjects that include dyspnea, cough, health-related quality of life, sleep quality, spirometry, a 6-minute walk test, and chest CT. All subjects, from both groups will also use the SPIREHEALTH Tag Device to measure their daily heart rate, respiratory rate, patient activity and calories. The group that is randomized to use the HHHFA device will be provided the HHHFA device at the baseline visit. Subjects will use the device during sleep for 6 weeks and both the HHHFA arm and the control arm will return for a 6 week follow up visit. At the 6 week follow up visit, participants will repeat all baseline evaluations. The study team will compare variables (e.g. FEV1) between baseline and 6-week visit in each treatment group. The study team will also compare changes in those variables over time between groups. To evaluate the effect of treatment between baseline and 6 weeks, the study team will use linear mixed effect models controlling for demographics and lung function.

Subjects who have been using the HHHFA device will be asked to stop using the device for the next 6 weeks. Both arms will then have a follow up phone call at the end of the 6 weeks (12 week follow up phone call visit). Subjects from both arms will continue to use the SPIREHEALTH and that data will be collected for both arms during that 6 week period.

Subjects who were previously randomized to the HHHFA arm will be asked, at the 6 week follow up visit, if they would be interested in participating in an optional sub-study that would allow them to start using the HHHFA device again, after their 12 week follow up phone call for an additional 36 weeks (for a total study involvement of 48 weeks) The subjects will have follow up phone call visits at 24 weeks, 36 weeks, and 48 weeks. Subjects who were randomized to the HHHFA device but do not want to keep using the device will be given the option of continuing to participate but only will the follow up phone call visits. Respiratory exacerbations information will be collected at these phone call visits.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis by health care provider
* Post-bronchodilator FEV1/FVC <0.7
* Post-bronchodilator FEV1%predicted <70%
* Chronic bronchitis, defined as chronic cough with daily sputum production
* ≥2 COPD exacerbations within the last year
* Smart phone

Exclusion Criteria:

* Obstructive sleep apnea and using positive airway pressure treatment
* Patients that use oxygen supplementation continuously (patients that use oxygen supplementation only at exertion will NOT be excluded)
* Any planned procedure that the PI believes would cause the subject to be ineligible.
* Unable to perform a spirometry, 6-minute walk test or chest CT
* Recent diagnosis (<4 weeks prior to study entry) of pneumonia, respiratory infection, COPD exacerbation, or acute bronchitis requiring antibiotics and new/increased dose of systemic corticosteroids
* Thoracic surgery or another procedure in the last six months that may result in instability of pulmonary status
* Recent medical or surgical history of upper airway disease that may interfere with intervention (e.g., sinus surgery, significant nasal polyps)
* Recent chest illness (trauma, pneumothorax etc).
* Basal skull surgery in the last 6 months
* Open skin ulcer or rash where the nasal cannula will be worn
* Tracheostomy or laryngectomy
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spyridon Fortis, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fortis S, Hoffman EA, Comellas AP. The Effect of Heated, Humidified High-Flow Air in COPD Patients With Chronic Bronchitis. Pulm Med. 2025 Dec 28;2025:8350741. doi: 10.1155/pm/8350741. eCollection 2025. PMID 41496867

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HHHFA Randomized Group | Control Group
Started | 8 | 3
Completed | 4 | 3
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HHHFA Randomized Group | Control Group | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 1 | 1 | 2
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 58 [56.5 to 63] | 61 [57.5 to 70] | 59 [56 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Sleep Quality Using the PSQI Questionnaire
Description: Pittsburgh Sleep Quality Index (PSQI) Questionnaires will be done at baseline and completion of study. This questionnaire will be used to collect information regarding the subject's usual sleep habits during the past month. PSQI: Pittsburgh Sleep Quality Index ranges from 0 to 21 with highest scores indicating worse sleep quality. Values presented here indicate the change between baseline and 6 weeks. Positive values indicate worse sleep quality at 6 weeks.
Time Frame: Baseline and 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HHHFA Randomized Group | Control Group
Number analyzed (Participants) | 4 | 3
score on a scale | -0.5 [-1.5 to 0.5] | 1 [-2.5 to 1]

2. Secondary Outcome: 6 Minute Walk
Description: Change in 6 minute walk distance. 6 min walk: distance covered during 6 min walk in meters. Greater values indicate better exercise capacity.
Time Frame: Baseline and 6 weeks
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | HHHFA Randomized Group | Control Group
Number analyzed (Participants) | 4 | 3
meters | 20 [-11 to 45] | 1.5 [-28 to 14]

3. Secondary Outcome: Health Related Quality of Life Change Using the CAT Questionnaire
Description: COPD Assessment Test (CAT) Questionnaires will be done at baseline and completion of study. This questionnaire will collect information regarding the subject's belief on the impact COPD is having on the wellbeing and daily life. CAT: COPD Assessment Test ranges from 0 to 40. Values presented here indicate the change between baseline and 6 weeks. Higher scores indicate worse quality of life due to COPD at 6 weeks.
Time Frame: Baseline and 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HHHFA Randomized Group | Control Group
Number analyzed (Participants) | 4 | 3
score on a scale | 0 [-0.25 to 1.25] | -7 [-9 to -3]

ADVERSE EVENTS:
Time Frame: From enrollment to 6 weeks.
Arm/Group | HHHFA Randomized Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT03959982/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT03959982/SAP_001.pdf